CLINICAL TRIAL: NCT07278479
Title: A Phase 1/2a Study to Assess Safety, Tolerability, and Efficacy of [212Pb]Pb-DOTAM-MAM279 in Patients With Small Cell Lung Cancer and Other DLL3 Expressing Solid Tumors
Brief Title: Study of [212Pb]Pb-DOTAM-MAM279 ([212Pb]Pb-MP0712) in Patients With Small Cell Lung Cancer and Other DLL3 Expressing Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Molecular Partners AG (Industry)
Collaborators: Orano Med LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MP0712-CP101
Record Dates: First submitted 2025-11-10; First posted 2025-12-12 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Large Cell Neuroendocrine Carcinoma; Large Cell Pulmonary Neuroendocrine Carcinoma of the Lung (LCNEC); Extrapulmonary Neuroendocrine Carcinoma (EP-NEC); Small Cell Lung Cancer (SCLC); Gastroenteropancreatic NEC (GEP NEC); NEC of the Bladder; Other DLL3 Expressing epNEC
Keywords: DARPin; Alpha Emitter; Pb203; Pb212; DLL3; Radioligand therapy (RLT); SCLC; Neuroendocrine cancer; [203Pb]Pb-DOTAM-MAM279; [212Pb]Pb-DOTAM-MAM279; EP-NEC; Lead 212; Lead 203; 203Pb; 212Pb
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Neuroendocrine

STUDY DESIGN:
Intervention Model Description: This is a phase 1/2a, multicenter, open-label study evaluating the safety, tolerability, and preliminary efficacy of [212Pb]Pb-DOTAM-MAM279 in patients with:
  * SCLC or LC NECs of the lung
  * epNECs
  The study is divided into two parts:
  * Part 1 (Phase 1): Dose escalation
  * Part 2 (Phase 2a): Dose expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [203Pb]Pb-DOTAM-MAM279/[212Pb]Pb-DOTAM-MAM279 (Experimental): Patients will receive [203Pb]Pb-DOTAM-MAM279 for Imaging/Dosimetry followed by [212Pb]Pb-DOTAM-MAM279 for treatment
  Interventions: Drug: [212Pb]Pb-MP0712; Other: [203Pb]Pb-MP0712

INTERVENTIONS:
Drug: [212Pb]Pb-MP0712 — Radioligand Therapy
  Other Names: [212Pb]Pb-DOTAM-MAM279
Other: [203Pb]Pb-MP0712 — Radioligand Imaging Agent
  Other Names: [203Pb]Pb-DOTAM-MAM279

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, dosimetry and preliminary efficacy of [212Pb]Pb-MP0712, in patients aged ≥18 years with Small Cell Lung Cancer and other locally advanced or metastatic DLL3 positive tumors.

DETAILED DESCRIPTION:
This is a phase I/IIa, open-label, multi-center study to evaluate the safety, tolerability, dosimetry, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of [212Pb]Pb-MP0712 in patients with SCLC and other advanced DLL3-expressing solid tumors. The study consists of a dose escalation part, followed by a dose expansion part. Once the recommended radioactive dose(s) [212Pb]Pb-MP0712 for further clinical evaluation are determined, the dose expansion part will further characterize the safety, tolerability, and preliminary anti-tumor activity of [212Pb]Pb-MP0712. The study will enable evaluation of the safety, dosimetry, PK, and imaging properties of [203Pb]Pb-MP0712.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years old
* Histologically or cytologically confirmed: I. advanced extensive or limited SCLC or LC NECs of the lung

  * SCLC (extensive stage, or limited stage) patients with progression or recurrence following at least two prior line of systemic platinum based therapy and immunotherapy or are not suitable or tolerating the standard of care treatment as second line of systemic therapy, or
  * LC NEC of the lung patients with progression or recurrence following at least one prior line of systemic therapy, or II. epNECs with progression or recurrence following at least one prior line of systemic therapy:
  * Gastroenteropancreatic NECs (GEPNEC), or
  * Cervical NECs, or
  * Bladder NECs, or
  * other epNECs with previously confirmed DLL3 expression by IHC.
  * Patients with prior DLL3-targeted therapy are allowed.
* For epNECs in Part 1 and Part 2 and SCLC or LC NECs of the lung in Part 2: DLL3-positivity by [203Pb]Pb-DOTAM-MAM279 SPECT/CT
* Radiographically documented disease progression or recurrence during or after the last line of systemic treatment therapy
* At least one measurable disease per RECIST v1.1.
* Adequate bone marrow reserve and organ function as demonstrated by complete blood count, and biochemistry in blood and urine at Screening
* Adequate blood counts: Hemoglobin ≥9 g/dL; Absolute neutrophil count (ANC) ≥1.5 × 10^9/L; Platelets ≥100 × 10^9/L; White blood cells (WBC) ≥2.5 x 10^9/L;
* Adequate hepatic function
* Adequate renal function: Calculated glomerular filtration rate (GFR) >60mL/min (using Cockroft-Gault formula).
* Patients with known central nervous system (CNS) metastasis will be eligible if they are clinically stable.

Key Exclusion Criteria:

* Uncontrolled intercurrent illness
* Patients who have not had resolution of all clinically significant toxic effects of prior systemic cancer therapy, surgery, or radiotherapy to Grade ≤1 (except for grade ≤2 alopecia, or stable grade 2 sensory neuropathy, according to the last CTCAE version).
* Active clinically significant cardiac disease
* Evidence of interstitial lung disease or active, non-infectious pneumonitis.
* History of other malignancy within the past 2 years with exceptions.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
To assess incidence and severity of safety events following administration of [212Pb]Pb-DOTAM-MAM279 | until 5 years after last dose
  Type, frequency and severity of adverse events (AEs), and serious adverse events (SAEs), Adverse events of special interest (AESI) and Dose Limiting Toxicities (DLT) using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE)
To assess dose modifications of [212Pb]Pb-DOTAM-MAM279 | until 5 years after last dose
  Frequency and duration of dose changes
To estimate the maximum tolerated dose (MTD) and/or to define the recommended phase 2 dose (RP2D) for SCLC/LCNEC of the lung and epNECs | Phase 1, from start of treatment to end of first cycle (day 1 - 28)
  Incidence of dose limiting toxicities
To evaluate the preliminary anti-tumor activity of [212Pb]Pb-DOTAM-MAM279 in the dose expansion part | Phase 2a only; 12 months
  Objective Response Rate (ORR) in the expansion phase
  ORR is defined as the percentage of patients with partial response (PR) or complete response (CR) as per RECIST v1.1

SECONDARY OUTCOMES:
To assess maximum concentration (Cmax) of [203Pb]Pb-DOTAM-MAM279 / [212Pb]Pb-DOTAM-MAM279 | up to 7 days following [203Pb]Pb-DOTAM-MAM279 administration; up to 14 days following [212Pb]Pb-DOTAM-MAM279 administration]
  Blood and serum samples will be drawn to determine maximum concentration (Cmax) of [203Pb]Pb-DOTAM-MAM279 / [212Pb]Pb-DOTAM-MAM279
To assess the area under the curve (AUC) from time 0 to the time of the last quantifiable concentration of [203Pb]Pb-DOTAM-MAM279 | up to 7 days following [203Pb]Pb-DOTAM-MAM279 administration; up to 14 days following [212Pb]Pb-DOTAM-MAM279 administration]
  Blood and serum samples will be drawn to determine AUC of [203Pb]Pb-DOTAM-MAM279 / [212Pb]Pb-DOTAM-MAM279
To assess half-live(s) (t½) of [203Pb]Pb-DOTAM-MAM279 / [212Pb]Pb-DOTAM-MAM279 | up to 7 days following [203Pb]Pb-DOTAM-MAM279 administration; up to 14 days following [212Pb]Pb-DOTAM-MAM279 administration]
  Blood and serum samples will be drawn to determine half-live(s) (t½) of [203Pb]Pb-DOTAM-MAM279 / [212Pb]Pb-DOTAM-MAM279
To assess the clearance (CL) of [203Pb]Pb-DOTAM-MAM279 / [212Pb]Pb-DOTAM-MAM279 | up to 7 days following [203Pb]Pb-DOTAM-MAM279 administration; up to 14 days following [212Pb]Pb-DOTAM-MAM279 administration]
  Blood and serum samples will be drawn to determine clearance (CL) of [203Pb]Pb-DOTAM-MAM279 / [212Pb]Pb-DOTAM-MAM279
To assess the volume of distribution (Vd) of [203Pb]Pb-DOTAM-MAM279 / [212Pb]Pb-DOTAM-MAM279 | up to 7 days following [203Pb]Pb-DOTAM-MAM279 administration; up to 14 days following [212Pb]Pb-DOTAM-MAM279 administration]
  Blood and serum samples will be drawn to determine the volume of distribution (Vd) of [203Pb]Pb-DOTAM-MAM279 / [212Pb]Pb-DOTAM-MAM279
To quantitatively predict radiation absorbed doses for therapeutic [212Pb]Pb-DOTAM-MAM279 from [203Pb]Pb-DOTAM-MAM279 | Phase 1; up to 7 days following [203Pb]Pb-DOTAM-MAM279 administration
  Estimation of [212Pb]Pb-DOTAM-MAM279 absorbed dose for healthy organs and tumor lesions based on dosimetry analysis of [203Pb]Pb-DOTAM-MAM279
To assess incidence and severity of safety events following administration of [203Pb]Pb-DOTAM-MAM279 | up to 10 days following [203Pb]Pb-DOTAM-MAM279 administration
  Type, frequency and severity of adverse events (AEs) and serious adverse events (SAEs) using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0
To evaluate PFS | Phase 2a only; 12 months
  Progression-Free Survival (PFS) determined as the time from C1D1 to the date of progression, defined as the first documented progression as per RECIST v1.1 or death for any cause
To evaluate DoR | Phase 2a only; 12 months
  Duration of response (DoR) in patients with a CR or PR from date of first date of response to the date of RECIST 1.1 progression or death
To evaluate DCR | Phase 2a only; 12 months
  Disease control rate (DCR) defined as the percentage of patients who have achieved CR, PR, or stable disease (SD)
To evaluate OS | Phase 2a only; approx. 5 years
  Overall survival (OS) defined as the time from C1D1 to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Nebraska Cancer Specialists, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided